CLINICAL TRIAL: NCT06259318
Title: Feasibility of Kanasina Gulabi, a Pilot Peer Support Intervention for Young Adults With Type 2 Diabetes in Mysore District, South India
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Public Health Research Institute of India (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0247; 2023-03-11-77 (Other: Public Health Research Institute of India)
Record Dates: First submitted 2024-01-29; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Type 2 Diabetes; Quality of Life; Depression; Stigma, Social; Behavior, Health
Keywords: Young Adult; India
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Social Stigma; Health Behavior

STUDY DESIGN:
Intervention Model Description: This study is a Hybrid Type 2 Effectiveness-Implementation Trial of a pilot, 2-arm, parallel-group, quasi-randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Kanasina Gulabi
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Kanasina Gulabi — Kanasina Gulabi is a theory-driven, educational-behavioral intervention designed to improve the quality of life and diabetes management among young adults living with type 2 diabetes in Mysore district, South India. In this intervention, young adults with type 2 diabetes were matched to non-specialist peer navigators -- trained young adult peers who were also managing type 2 diabetes -- and developed action plans to improve their physical and mental health outcomes. Intervention components included group education, mindfulness activities, self care activity tracking, and phone follow-ups to address knowledge gaps and misinformation about type 2 diabetes, build self-efficacy for type 2 diabetes-related self care activities, and provide emotional support for diabetes management.
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate a pilot peer support intervention, entitled "Kanasina Gulabi" (Translation "My Dream Rose" in Kannada), designed to improve quality of life and diabetes management among young adults living with type 2 diabetes. The intervention, delivered by non-specialist providers - trained young adult peer navigators who are also managing type 2 diabetes - is expected to improve physical and mental health outcomes among participants. The sample includes young adults aged 18-40 with a diagnosis of type 2 diabetes in Mysore district, South India. Participants were quasi-randomly allocated to the intervention or control group. With the support of their peer navigators, intervention participants will develop action plans to improve their physical and mental health outcomes. This study plans to assess the feasibility, acceptability, and preliminary effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 - 40 years old
* self-reported to have type 2 diabetes
* living in Mysore district
* able to speak English or Kannada
* and able to access a cellular phone during the study period

Exclusion Criteria:

* pregnant
* living with a serious medical or psychological disorder that would impede study procedure

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Reach | Week 0 - 5, Week 12
  The absolute number, proportion, and representativeness of individuals who are willing to participate in the quasi-experimental study for Kanasina Gulabi.
Glycemic Control | Week 0, Week 12
  Percentage of measured hemoglobin A1c (HbA1c) that represents average blood sugar levels over the past 3 months, used to measure diabetes management and glycemic control.
Diabetes Knowledge | Week 0, Week 5, Week 12
  Diabetes Knowledge Questionnaire (DKQ-24). 24 self-report items to assess overall diabetes knowledge. Responses are measured as true, false, or don't know. One composite score is calculated (range: 0 - 24); higher scores reflect better diabetes knowledge.
Diabetes Distress | Week 0, Week 5, Week 12
  Type 2 Diabetes Distress Assessment System (T2-DDAS). 8 self-report items to assess diabetes-related emotional distress in adults with type 2 diabetes. Responses are endorsed on a 5-point scale and refer to the past month. One composite mean score is calculated (range: 0 - 5); higher scores reflect more diabetes distress.
Diabetes-Related Stigma | Week 0, Week 5, Week 12
  Type 2 Diabetes Stigma Assessment Scale (DSAS-2). 19 self-report items to assess perceived and experienced stigma for adults with type 2 diabetes. Responses are endorsed on a 5-point scale and refer to the past two weeks. One composite score is calculated (range: 19 - 95); higher scores reflect more experiences of stigma.
Depressive Symptoms | Week 0, Week 5, Week 12
  Patient Health Questionnaire (PHQ-9). 9 self-report items to screen for depression and assess degree of severity. Responses are endorsed on a 4-point scale and refer to the past two weeks. One composite score is calculated (range: 0 - 27); higher scores reflect more depressive symptoms.
Optimism | Week 0, Week 5, Week 12
  Revised Life Orientation Test (LOT-R). 10 self-report items to measure positive and negative expectations strongly linked to the future. Responses are endorsed on a 5-point scale. One composite score is calculated (range: 0 - 24); higher scores reflect higher dispositional optimism.

CONTACTS AND LOCATIONS:
Overall Officials: Eve S Puffer, PhD, Principal Investigator — Duke University; Sumedha Ariely, PhD, Principal Investigator — Duke University
Locations (1):
- Public Health Research Institute of India, Mysore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No